CLINICAL TRIAL: NCT00000158
Title: Macular Photocoagulation Study (MPS)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-60
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-06

CONDITIONS: Choroidal Neovascularization; Macular Degeneration; Histoplasmosis
Keywords: photocoagulation; argon blue-green laser; krypton red laser
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration; Histoplasmosis

INTERVENTIONS:
Procedure: Argon Blue-Green Laser Photocoagulation

SUMMARY:
To evaluate laser treatment of choroidal neovascularization (CNV) through randomized, controlled clinical trials. The Macular Photocoagulation Study (MPS) consisted of three sets of randomized, controlled clinical trials. Change in best-corrected visual acuity from baseline was the primary outcome for all MPS trials. Other measures of vision are evaluated in each set of trials. The purpose of each is described below.

Argon Study: To determine whether argon blue-green laser photocoagulation of leaking abnormal blood vessels in choroidal neovascular membranes outside the fovea (200 to 2,500 microns from the center of the foveal avascular zone [FAZ]) is of benefit in preventing or delaying loss of central vision in patients with age-related (senile) macular degeneration (AMD), presumed ocular histoplasmosis (POH), and idiopathic neovascular membranes (INVM). A separate trial was conducted for each of the three underlying conditions.

Krypton Study: To determine whether krypton red laser photocoagulation of choroidal neovascular lesions with the posterior border 1 to 199 microns from the center of the FAZ is of benefit in preventing or delaying large losses of visual acuity in patients with AMD, POH, and INVM. A separate trial was conducted for each of the three underlying conditions.

Foveal Study: To determine whether laser photocoagulation is of benefit in preventing or delaying further visual acuity loss in patients with new (never treated) or recurrent (previously treated with laser photocoagulation) choroidal neovascularization under the center of the FAZ. Two separate trials, one for each type of lesion, were carried out.

DETAILED DESCRIPTION:
In each randomized trial conducted by the MPS Group, focal laser photocoagulation was compared to observation without treatment. Patients were assigned to laser treatment or to observation with equal probability. The first set of MPS randomized trials, the Argon Study, focused on the effectiveness of photocoagulation with argon blue-green laser in eyes with discrete extrafoveal choroidal neovascularization. The study investigators, who began recruiting patients in 1979, estimated that 550 patients with AMD and 750 with POH would be required. Follow-up was to continue for 5 years to determine whether argon laser photocoagulation treatment could prevent or delay visual acuity loss in these patients.

After the initiation of the Argon Study, a new krypton red laser became available. The new wavelength offered theoretical advantages over the argon laser for treating CNV that extended inside the FAZ of the macula. The Krypton Study design was analogous to the Argon Study, with the investigation of three underlying conditions, except that CNV was closer to the FAZ center.

The third set of MPS clinical trials, the Foveal Study, was designed to determine whether laser photocoagulation was effective for delaying or preventing further visual acuity loss in AMD patients who have subfoveal CNV. Among patients assigned to laser treatment in the Foveal Study, argon laser treatment was compared with krypton red laser treatment of these lesions. The investigators originally projected that about 350 patients would be required for each clinical trial of the Foveal Study.

ELIGIBILITY:
Common Eligibility Criteria for the Argon, Krypton, and Foveal Studies:

To be eligible, men and women must have been experiencing visual symptoms attributable to the macular lesion, such as decreased visual acuity or Amsler grid distortion, at the time of entry into the study. They also must have had visible, well-demarcated hyperfluorescence characteristic of classic choroidal neovascularization on fluorescein angiography. AMD patients were 50 years of age or older and had drusen visible in the macula of at least one eye. POH patients were at least 18 years old and had at least one characteristic histo spot in one or both eyes. INVM patients were at least 18 years old and had no evidence of AMD, POH, angioid streaks, high myopia, diabetic retinopathy, or any other condition that could be the cause of the neovascularization. In particular, INVM patients had neither drusen greater than MPS Standard Photograph No. 1.1 nor histo spots in either eye.

Additional Patient Eligibility Criteria for the Argon Study:

Each patient had a visible serous detachment of the sensory retina with a diffuse area of leakage, discrete choroidal neovascularization outside the fovea (200-2,500 microns from the center of the FAZ), and visual acuity of 20/100 or better in the study eye.

Additional Patient Eligibility Criteria for the Krypton Study:

All patients had a neovascular lesion consisting of neovascularization and possibly blood and/or pigment that extended into the FAZ. The posterior border of CNV could extend as close as 1 micron to the FAZ center. Visual acuity of the study eye was 20/400 or better.

Additional Patient Eligibility Criteria for the Foveal Study:

Only patients with AMD were eligible for this study. Fluorescein angiography of the eligible eye had to show evidence of a leaking choroidal neovascular membrane, some part of which extended under the center of the FAZ, or a neovascular lesion consisting of an old laser treatment scar and contiguous leaking neovascularization within 150 microns of the center of the FAZ. New, never-treated subfoveal lesions were less than four disc areas in size. Recurrent lesions were less than six disc areas in size, including the old treatment scar and new neovascularization. Best-corrected visual acuity was no better than 20/40 and no worse than 20/320.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1979-02

REFERENCES:
- [Background] Changing the protocol: a case report from the Macular Photocoagulation Study. Macular Photocoagulation Study Group. Control Clin Trials. 1984 Sep;5(3):203-16. doi: 10.1016/0197-2456(84)90024-2. PMID 6488805
- [Background] Hillis A, Maguire M, Hawkins BS, Newhouse MM. The Markov process as a general method for nonparametric analysis of right-censored medical data. J Chronic Dis. 1986;39(8):595-604. doi: 10.1016/0021-9681(86)90184-0. PMID 3525597
- [Background] Blackhurst DW, Maguire MG. Reproducibility of refraction and visual acuity measurement under a standard protocol. The Macular Photocoagulation Study Group. Retina. 1989;9(3):163-9. PMID 2480626
- [Background] Hawkins BS, Prior MJ, Fisher MR, Blackhurst DW. Relationship between rate of patient enrollment and quality of clinical center performance in two multicenter trials in ophthalmology. Control Clin Trials. 1990 Oct;11(5):374-94. doi: 10.1016/0197-2456(90)90177-4. PMID 1963130
- [Background] Argon laser photocoagulation for senile macular degeneration. Results of a randomized clinical trial. Arch Ophthalmol. 1982 Jun;100(6):912-8. doi: 10.1001/archopht.1982.01030030920003. PMID 7046707
- [Background] Argon laser photocoagulation for ocular histoplasmosis. Results of a randomized clinical trial. Arch Ophthalmol. 1983 Sep;101(9):1347-57. doi: 10.1001/archopht.1983.01040020349002. PMID 6193771
- [Background] Argon laser photocoagulation for idiopathic neovascularization. Results of a randomized clinical trial. Arch Ophthalmol. 1983 Sep;101(9):1358-61. doi: 10.1001/archopht.1983.01040020360003. PMID 6193772
- [Background] Fine SL. Early detection of extrafoveal neovascular membranes by daily central field evaluation. Ophthalmology. 1985 May;92(5):603-9. doi: 10.1016/s0161-6420(85)33995-7. PMID 2409502
- [Background] Recurrent choroidal neovascularization after argon laser photocoagulation for neovascular maculopathy. Macular Photocoagulation Study Group. Arch Ophthalmol. 1986 Apr;104(4):503-12. doi: 10.1001/archopht.1986.01050160059012. PMID 2420315
- [Background] Argon laser photocoagulation for neovascular maculopathy. Three-year results from randomized clinical trials. Macular Photocoagulation Study Group. Arch Ophthalmol. 1986 May;104(5):694-701. PMID 2423061
- [Background] Krypton laser photocoagulation for neovascular lesions of ocular histoplasmosis. Results of a randomized clinical trial. Macular Photocoagulation Study Group. Arch Ophthalmol. 1987 Nov;105(11):1499-507. doi: 10.1001/archopht.1987.01060110045029. PMID 2445326
- [Background] Chamberlin JA, Bressler NM, Bressler SB, Elman MJ, Murphy RP, Flood TP, Hawkins BS, Maguire MG, Fine SL. The use of fundus photographs and fluorescein angiograms in the identification and treatment of choroidal neovascularization in the Macular Photocoagulation Study. The Macular Photocoagulation Study Group. Ophthalmology. 1989 Oct;96(10):1526-34. doi: 10.1016/s0161-6420(89)32707-2. PMID 2479899
- [Background] Persistent and recurrent neovascularization after krypton laser photocoagulation for neovascular lesions of ocular histoplasmosis. Macular Photocoagulation Study Group. Arch Ophthalmol. 1989 Mar;107(3):344-52. doi: 10.1001/archopht.1989.01070010354023. PMID 2466454
- [Background] Krypton laser photocoagulation for neovascular lesions of age-related macular degeneration. Results of a randomized clinical trial. Macular Photocoagulation Study Group. Arch Ophthalmol. 1990 Jun;108(6):816-24. doi: 10.1001/archopht.1990.01070080058036. PMID 1693496
- [Background] Persistent and recurrent neovascularization after krypton laser photocoagulation for neovascular lesions of age-related macular degeneration. Macular Photocoagulation Study Group. Arch Ophthalmol. 1990 Jun;108(6):825-31. doi: 10.1001/archopht.1990.01070080067037. PMID 1693497
- [Background] Krypton laser photocoagulation for idiopathic neovascular lesions. Results of a randomized clinical trial. Macular Photocoagulation Study Group. Arch Ophthalmol. 1990 Jun;108(6):832-7. PMID 1693498
- [Background] Bressler SB, Maguire MG, Bressler NM, Fine SL. Relationship of drusen and abnormalities of the retinal pigment epithelium to the prognosis of neovascular macular degeneration. The Macular Photocoagulation Study Group. Arch Ophthalmol. 1990 Oct;108(10):1442-7. doi: 10.1001/archopht.1990.01070120090035. PMID 1699513
- [Background] Bressler NM, Bressler SB, Alexander J, Javornik N, Fine SL, Murphy RP. Loculated fluid. A previously undescribed fluorescein angiographic finding in choroidal neovascularization associated with macular degeneration. Macular Photocoagulation Study Reading Center. Arch Ophthalmol. 1991 Feb;109(2):211-5. doi: 10.1001/archopht.1991.01080020057043. PMID 1704212
- [Background] Argon laser photocoagulation for neovascular maculopathy. Five-year results from randomized clinical trials. Macular Photocoagulation Study Group. Arch Ophthalmol. 1991 Aug;109(8):1109-14. PMID 1714270
- [Background] Laser photocoagulation of subfoveal recurrent neovascular lesions in age-related macular degeneration. Results of a randomized clinical trial. Macular Photocoagulation Study Group. Arch Ophthalmol. 1991 Sep;109(9):1232-41. doi: 10.1001/archopht.1991.01080090056026. PMID 1718251
- [Background] Subfoveal neovascular lesions in age-related macular degeneration. Guidelines for evaluation and treatment in the macular photocoagulation study. Macular Photocoagulation Study Group. Arch Ophthalmol. 1991 Sep;109(9):1242-57. PMID 1718252
- [Background] Birch DG, Anderson JL, Fish GE, Jost BF. Pattern-reversal electroretinographic acuity in untreated eyes with subfoveal neovascular membranes. Invest Ophthalmol Vis Sci. 1992 Jun;33(7):2097-104. PMID 1376721
- [Background] Orr PR, Blackhurst DW, Hawkins BS. Patient and clinic factors predictive of missed visits and inactive status in a multicenter clinical trial. The Macular Photocoagulation Study Group. Control Clin Trials. 1992 Feb;13(1):40-9. doi: 10.1016/0197-2456(92)90028-x. PMID 1315662
- [Background] Birch DG, Anderson JL, Fish GE, Jost BF. Pattern-reversal electroretinographic follow-up of laser photocoagulation for subfoveal neovascular lesions in age-related macular degeneration. Am J Ophthalmol. 1993 Aug 15;116(2):148-55. doi: 10.1016/s0002-9394(14)71278-4. PMID 8352298
- [Background] Fine SL; The case for treating subfoveal neovascularization in patients with age-related macular degeneration, Franklin RM (ed): Retina and Vitreous., Proceedings of the Symposium on Retina and Vitreous, New Orleans Academy of Ophthalmology, New York, Kugler Publications 1993:29-30
- [Background] Five-year follow-up of fellow eyes of patients with age-related macular degeneration and unilateral extrafoveal choroidal neovascularization. Macular Photocoagulation Study Group. Arch Ophthalmol. 1993 Sep;111(9):1189-99. doi: 10.1001/archopht.1993.01090090041018. PMID 7689826
- [Background] Laser photocoagulation of subfoveal neovascular lesions of age-related macular degeneration. Updated findings from two clinical trials. Macular Photocoagulation Study Group. Arch Ophthalmol. 1993 Sep;111(9):1200-9. doi: 10.1001/archopht.1993.01090090052019. PMID 7689827
- [Background] Visual outcome after laser photocoagulation for subfoveal choroidal neovascularization secondary to age-related macular degeneration. The influence of initial lesion size and initial visual acuity. Macular Photocoagulation Study Group. Arch Ophthalmol. 1994 Apr;112(4):480-8. doi: 10.1001/archopht.1994.01090160056023. PMID 7512334
- [Background] Persistent and recurrent neovascularization after laser photocoagulation for subfoveal choroidal neovascularization of age-related macular degeneration. Macular Photocoagulation Study Group. Arch Ophthalmol. 1994 Apr;112(4):489-99. doi: 10.1001/archopht.1994.01090160065024. PMID 7512335
- [Background] Laser photocoagulation for juxtafoveal choroidal neovascularization. Five-year results from randomized clinical trials. Macular Photocoagulation Study Group. Arch Ophthalmol. 1994 Apr;112(4):500-9. PMID 7512336
- [Background] Evaluation of argon green vs krypton red laser for photocoagulation of subfoveal choroidal neovascularization in the macular photocoagulation study. Macular Photocoagulation Study (MPS) Group. Arch Ophthalmol. 1994 Sep;112(9):1176-84. doi: 10.1001/archopht.1994.01090210060017. PMID 7522004
- [Background] Laser photocoagulation for neovascular lesions nasal to the fovea. Results from clinical trials for lesions secondary to ocular histoplasmosis or idiopathic causes. Macular Photocoagulation Study Group. Arch Ophthalmol. 1995 Jan;113(1):56-61. PMID 7529993
- [Background] The influence of treatment extent on the visual acuity of eyes treated with Krypton laser for juxtafoveal choroidal neovascularization. Macular Photocoagulation Study Group. Arch Ophthalmol. 1995 Feb;113(2):190-4. doi: 10.1001/archopht.1995.01100020074032. PMID 7532395
- [Background] Occult choroidal neovascularization. Influence on visual outcome in patients with age-related macular degeneration. Macular Photocoagulation Study Group. Arch Ophthalmol. 1996 Apr;114(4):400-12. PMID 8602776
- [Background] Five-year follow-up of fellow eyes of individuals with ocular histoplasmosis and unilateral extrafoveal or juxtafoveal choroidal neovascularization. Macular Photocoagulation Study Group. Arch Ophthalmol. 1996 Jun;114(6):677-88. doi: 10.1001/archopht.1996.01100130669006. PMID 8639078
- [Background] Risk factors for choroidal neovascularization in the second eye of patients with juxtafoveal or subfoveal choroidal neovascularization secondary to age-related macular degeneration. Macular Photocoagulation Study Group. Arch Ophthalmol. 1997 Jun;115(6):741-7. doi: 10.1001/archopht.1997.01100150743009. PMID 9194725
- [Derived] Hawkins BS, Bressler NM, Reynolds SM. Visual acuity outcomes among sham vs no-treatment controls from randomized trials. Arch Ophthalmol. 2009 Jun;127(6):725-31. doi: 10.1001/archophthalmol.2009.101. PMID 19506188